CLINICAL TRIAL: NCT05408364
Title: Clinical and Microbiological Evaluation of Probiotics as an Adjunct to Initial Periodontal Treatment in Chronic Periodontitis
Brief Title: Probiotics Effects to Initial Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAR-2011-03-30-24
Record Dates: First submitted 2022-05-16; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2011-03

CONDITIONS: Chronic Periodontitis
Keywords: bifidobacterium; chronic periodontitis; dental scaling; probiotic; root planing
MeSH Terms: conditions — Chronic Periodontitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Individuals and doctor were blinded to the study groups allocation. Before statistical analysis, the blind study coordinator broke the code to allocate the indivuals to the groups.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Natural yoghurt (Placebo Comparator): SRP+nature yogurt (Danone® yogurt, Luleburgaz, Türkiye)
  Interventions: Dietary Supplement: probiotic or natural yoghurt; Procedure: SRP
- Probiotic yoghurt (Experimental): SRP+probiotic containing yogurt (Danone Activia® Plain, Luleburgaz, Türkiye)
  Interventions: Dietary Supplement: probiotic or natural yoghurt; Procedure: SRP

INTERVENTIONS:
Dietary Supplement: probiotic or natural yoghurt — Bifidobacterium animalis subsp. lactis DN-173010 containing probiotic yoghurt
Procedure: SRP — Scalling and root planing

SUMMARY:
The aim of this study is to evaluate the clinical and microbiological effects of Bifidobacterium animalis subsp. lactis DN-173010 containing yoghurt as an adjunct to mechanical periodontal treatment.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the clinical and microbiological effects of Bifidobacterium animalis subsp. lactis DN-173010 containing yoghurt as an adjunct to mechanical periodontal treatment.

Thirty chronic periodontitis patients were randomized into 2 groups. As adjunctive to MPT, Group 1 consumed 2×108 CFU/day of Bifidobacterium animalis subsp. lactis DN-173010 containing probiotic yoghurt while Group 2 natural yoghurt once daily for 28 days. Subgingival plaque samples were obtained from 2 periodontal sites with probing pocket depth (PPD) of 4≤PPD<7 mm via paper-points at baseline, 28th day, 3rd month. Samples were cultured to evaluate total viable count (TVC), the proportions of obligate anaerobes (OA) and Bifidobacterium species (B) (TVC%). The full-mouth recorded clinical parameters were plaque index, gingival index, PPD, bleeding on probing, and clinical attachment level.

ELIGIBILITY:
Inclusion Criteria:

* chronic periodontitis patients with radiographically detected horizontal bone loss
* the presence of at least 2 teeth with one approximal site with a probing pocket depth (PPD) of 4≤SD<7 mm (5-7 mm) and a GI of ≥2 mm in each quadrant,
* previously untreated periodontitis, systemically healthy

Exclusion Criteria:

* Systemic diseases
* Antibiotics and anti-inflammatory drugs within 3 months before the study
* Untreated caries lesions or local retention factors
* Allergic reactions to lactose or fermented milk products
* Previous probiotic supplements in diet
* Smoking
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Probing Depth | 28 days
  Probing depth is defined as the distance from the free gingival margin to the bottom of the periodontal pocket.

SECONDARY OUTCOMES:
Gingival Index | 28 days
  Each of the buccal, mesial, lingual and distal surfaces of the gingival tissues is given a score of 0-3. (0 = Normal gingiva. 1 = Mild inflammation - slight change in color, slight edema. No bleeding on probing. 2. Moderate inflammation - redness, edema and glazing. Bleeding on probing. 3. Severe inflammation -marked redness and edema.)
Plaque Index | 28 days
  Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3. (0 = No plaque in the gingival area. 1 = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface. 2 = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye. 3 = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface. Tendency to spontaneous bleeding.)
Bleeding on probing | 28 days
  Bleeding on probing is defined as presence of bleeding from gingival sulcus during the probing of this area via periodontal probe.
Clinical attachment level | 28 days
  The distance from the cementoenamel junction to the bottom of the periodontal pocket.
microbiological parameters | 28 days
  The number of obligate anaerobic bacteria and Bifidobacterium anaerobes

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Kuru, Prof. Dr., Study Director — Marmara University, Faculty of Dentistry, Department of Periodontology; Hafize Öztürk Özener, Dr., Principal Investigator — Marmara University, Faculty of Dentistry, Department of Periodontology
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)